CLINICAL TRIAL: NCT02426229
Title: Safety & Suitability of Dabigatran to Inhibit Thrombin in Scleroderma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1R21AR065089-01A1 (NIH); 1R21AR065089-01A1 (NIH)
Record Dates: First submitted 2015-03-04; First posted 2015-04-24 (Estimated); Last update posted 2018-07-13 (Actual); Status verified 2018-07

CONDITIONS: Scleroderma; Interstitial Lung Disease
Keywords: SSc; systemic sclerosis; cutaneous systemic sclerosis
MeSH Terms: conditions — Scleroderma, Diffuse; Lung Diseases, Interstitial; Scleroderma, Systemic | interventions — Dabigatran

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- dabigatran 75mg (Experimental): dabigatran etexilate 75mg orally twice daily for 6 months
  Interventions: Drug: dabigatran etexilate

INTERVENTIONS:
Drug: dabigatran etexilate — dabigatran etexilate 75mg orally twice a day for 6 months
  Other Names: Dabigatran; Pradaxa

SUMMARY:
This study evaluates if dabigatran etexilate is safe for use in patients with Scleroderma and Interstitial Lung Disease. All patients will receive 75mg of dabigatran etexilate twice a day for 6 months.

DETAILED DESCRIPTION:
Skin and pulmonary fibrosis result in substantial morbidity in scleroderma (SSc). Furthermore, interstitial lung disease (ILD) culminating in pulmonary fibrosis is a major cause of death among scleroderma patients. Studies implicate the coagulation system, most notably the serine protease thrombin, in the pathogenesis of SSc-ILD. Thrombin can transform normal lung fibroblasts to a scleroderma fibroblast phenotype. Dabigatran etexilate is a selective thrombin inhibitor which is FDA-approved for the prevention of thromboembolic complications in patients with atrial fibrillation. Dabigatran etexilate needs to be studied as a potential anti-fibrotic agent for the treatment of SSc-ILD. This study is designed to see if dabigatran etexilate is safe for use in patients with scleroderma. If so, the long term goal of this study is to determine whether or not the fundamental results will translate to a potential clinical intervention for SSc-ILD which can be tested in a future randomized control trial.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤ 70 years
* All patients must fulfill the ACR/EULAR criteria for SSc. Patients may have limited (cutaneous thickening distal, but not proximal to elbows and knees, with or without facial involvement) or diffuse (cutaneous thickening proximal to elbows and knees, often involving the chest or abdomen) cutaneous SSc, or systemic sclerosis sine scleroderma
* SSc for less than 7 years, with onset defined as the date of the first non-Raynaud phenomenon manifestation.
* All patients must have interstitial lung disease defined by any ground glass on HRCT and >20% involvement of HRCT by pulmonary fibrosis and/or FVC <70% predicted

Exclusion Criteria:

* Inability to sign consent
* Currently enrolled in another clinical trial
* FVC < 40% predicted and/or DLCO (corrected for hemoglobin) < 30% of predicted (suggesting severe probably irreparable disease)
* Other serious concomitant medical illnesses (e.g., cancer) limiting life expectancy to <1 year at time of enrollment
* FEV1/FVC ratio < 65% (suggesting obstructive disease)
* Clinically significant pulmonary hypertension requiring treatment, based on the clinician's judgment.
* Smoking of cigars, pipes or cigarettes within 3 months prior to and during enrollment
* Clinically significant abnormalities on chest x-ray other than interstitial lung disease (e.g., lung mass, evidence of active pulmonary infection, emphysema)
* Use of prednisone (or equivalent) in doses > 10 mg daily within 3 months prior to and during enrollment
* Use of colchicine, D-penicillamine, cyclophosphamide, mycophenolate mofetil, azathioprine, endothelin receptor antagonists, phosphodiesterase type-5 inhibitors, prostanoids, tyrosine kinase inhibitors, sirolimus, rituximab, perfinidone or other "disease modifying medications" within 3 months prior to and during enrollment
* Pregnancy or lack of use of birth control method in women of childbearing age or lactating
* Liver disease or increased baseline liver enzyme levels (ALT >3 x upper limit of normal)
* Use of CYP450 inhibitors/inducers
* Hemoglobin < 10g/L
* If of child bearing potential, unwillingness to employ a reliable means of contraception (condom, abstinence, IUD, tubal ligation, vasectomy)
* Active infection
* Creatinine clearance <30 ml/min
* Post transplantation
* Active medical and psychiatric conditions which the investigator may consider would interfere with the subject's treatment, assessment, or compliance with the protocol
* Anticoagulation-related exclusions include:

  1. Current anticoagulation therapy with warfarin
  2. Increased risk of bleeding (e.g., uncorrectable inherited or acquired bleeding disorder)
  3. Platelet count <100,000/cmm or hematocrit <30% or > 55%
  4. History of severe gastrointestinal bleeding within 6 months of screening
  5. Known gastric antral vascular ectasia (GAVE) or gastric/intestinal arterial-venous malformations (AVMs)
  6. History of CVA within 6 months of screening
  7. History of risks of falls as judged by the PI
  8. Surgery or major trauma within the past 30 days
  9. Any condition that, in the determination of the PI, is likely to require anticoagulation therapy during the study
  10. Clopidogrel, prasugrel or other anti-platelet therapy within 6 months of screening
  11. Aspirin therapy >325 mg daily
  12. Therapy with other thrombin inhibitors

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-02; Primary Completion 2018-06 (Actual); Study Completion 2018-06-21 (Actual)

PRIMARY OUTCOMES:
Composite: Safety of dabigatran patients with scleroderma interstitial lung disease. (complete blood counts, comprehensive metabolic profile, and coagulation studies). | Up to 6 months
  Subjects taking dabigatran will undergo monthly complete blood counts (white blood cell count, hemoglobin, hematocrit, platelet), comprehensive metabolic profile (sodium, potassium, chloride, bicarbonate, BUN, creatinine, glucose, total bilirubin, AST, ALT, alkaline phosphatase, protein and albumin), and coagulation studies (prothrombin time, partial thromboplastin time and thrombin time). Women of child-bearing age will be required to have a urine pregnancy test monthly while receiving dabigatran.

SECONDARY OUTCOMES:
Composite: Preliminary estimate of efficacy of dabigatran in scleroderma. (skin score and dermal fibroblast biology) | Up to 6 months
  We will also include investigations of scleroderma skin (skin score and dermal fibroblast biology) together with studies of scleroderma lung fibroblasts, to obtain preliminary estimates of the effectiveness of dabigatran as a potential disease modifying drug for patients with SSc-ILD.

CONTACTS AND LOCATIONS:
Overall Officials: Richard M Silver, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

REFERENCES:
- [Background] Bogatkevich GS, Ludwicka-Bradley A, Silver RM. Dabigatran, a direct thrombin inhibitor, demonstrates antifibrotic effects on lung fibroblasts. Arthritis Rheum. 2009 Nov;60(11):3455-64. doi: 10.1002/art.24935. PMID 19877031
- [Derived] Bogatkevich GS, Huggins TJ, Ismail AA, Atanelishvili I, Silver RM. Anti-fibrotic effects of thrombin inhibition in systemic sclerosis-associated interstitial lung disease: Proof of concept. J Scleroderma Relat Disord. 2025 Feb 24:23971983241311625. doi: 10.1177/23971983241311625. Online ahead of print. PMID 40013233